CLINICAL TRIAL: NCT01831492
Title: Effects of Dietary Zeolite + Dolomite on Performance, Exercise-induced Acidosis, Oxidative Stress, Inflammation and Intestinal Barrier Dysfunction in Trained People
Brief Title: Effects of Zeolite + Dolomite on Performance and Acidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Pricipal Investigator, Green Beat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 25-217 ex 12/13; PSS (Other Grant/Funding Number: Panaceo International Active Mineral Production GmbH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Acidosis; Oxidative Stress; Inflammation
Keywords: performance; acidosis; oxidative stress; inflammation; oxygen uptake
MeSH Terms: conditions — Acidosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zeolite + dolomite (Active Comparator): 28 trained subjects receive encapsulated zeolite + dolomite
  Interventions: Device: zeolite + dolomite
- cellulose (Placebo Comparator): 28 trained subjects receive encapsulated micro-crystalline cellulose
  Interventions: Device: cellulose

INTERVENTIONS:
Device: zeolite + dolomite — Given for 12 weeks, after a 4 weeks wash- out of all supplements/drugs
  Other Names: Panaceo Sport
  Arms: zeolite + dolomite
Device: cellulose — given for 14 weeks
  Other Names: placebo
  Arms: cellulose

SUMMARY:
Purpose:

This study investigates the effects of dietary zeolite + dolomite on performance, exercise-induced acidosis, oxidative stress, inflammation and intestinal barrier dysfunction in trained people.

Hypotheses (H1):

Zeolite + dolomite increase performance in an ergometer step test Zeolite + dolomite reduce exercise-induced acidosis Zeolite + dolomite reduce oxidative stress Zeolite + dolomite reduce inflammation Zeolite + dolomite improve intestinal barrier dysfunction

DETAILED DESCRIPTION:
The application of adequate nutraceuticals for sporty people´s performance and health becomes more and more interesting for athletes and their carers. There are also great opportunities for product providers in this field to act commercially profitable.

Beside the main goal - to achieve improved performance - modern sport nutraceuticals should support immunity of athletes in all corners of health. One of the most interesting approaches in this field is to promote performance and health via dietary zeolites. Zeolites are synthetic microporous crystals containing AIO4 and SiO4 tetrahedrons. It is hypothesized that in human body these silicates act as gut-located adsorbents of chymus molecules or as ion-exchangers, catalysts, detergent builders or antidiarrheic agents (1, 2, 3, 4). These - mainly physical - effects of dietary used zeolite might also influence the chief issues of modern sport nutrition: performance, acidosis, oxidative stress, inflammation, gastrointestinal complaints and associated impacts on immunity and health.

The investigators hypothesize that the physical effects of zeolite affect the metabolism in the gut and exert systemic physiological/biochemical benefits in regard to human´s exercise performance, redox biology, inflammatory processes, acid-base balance, and even intestinal barrier integrity/function. All these postulated benefits would have tremendous impact on sports performance. However, up to date no clinical study is reported on PubMed that addresses these chief aims of sport nutrition in the context of zeolite supplementation.

GOALS

This protocol describes a study that investigates the effects of dietary zeolite + dolomite (Product name: "PANACEO SPORT") on performance, exercise-induced (acute or chronically) acidosis, oxidative stress, inflammation and intestinal barrier dysfunction. This is a randomized, placebo-controlled, double-blinded, parallel-grouped study design. In detail, the investigators want to assess the effects of dietary zeolite + dolomite (the commercially available product "PANACEO-SPORT") on:

1. Aerobic performance capability and maximum oxygen uptake (primary outcome)
2. Lactate kinetics and maximum lactate concentrations in blood (secondary outcome)
3. Oxidative stress (OS)/redox biology and inflammation (tertiary outcome)
4. Intestinal barrier integrity and endotoxemia (quaternary outcome) The investigators hypothesize that the intake of the product will beneficially influence outcomes 1-4 (H1-hypotheses 1-4: "Supplementation will influence...").

   MERITS of this study Data of this project will provide knowledge regarding the effects of zeolite and dolomite on aerobic performance, lactate kinetics, redox biology, inflammation and integrity of intestinal barrier. Results will help us to identify how to support chronically exercising people to optimize their performance and health.

   METHODS
   * Subjects: 56 healthy men, non-professional but homogeneously trained (>50ml/kg/min) triathletes and/or cyclists and/or dual athletes, non-smokers, 20-50 yrs, comparable body fat content (<20%) and psycho-physical stress profile, non-medicated, preventive

   medical check-up and actual proofed eligibility to conduct sports, pre-selection via telephone interviews.
   * Design: randomized, double-blinded, placebo-controlled, 2-arm parallel-group design. One arm is the placebo group, the second arm receives zeolite + dolomite ("PANACEO-SPORT"). After a wash-out of 4wk from any food supplements, also from specific dietetic and drug treatment, a period of 12wk with supplementation or placebo follows. At 0wk, 4wk and 12wk we conduct performance diagnostics. At 0wk and 12wk we collect blood and stool.
   * Treatment: Subjects receive 6 capsules per day of zeolite + dolomite ("PANACEO-SPORT") or placebo capsules with identical appearance. Subjects will be instructed to consume 3 capsules with the first meal of the day and 3 capsules with the last meal of the day. We recommend to dispense one box per subject and to produce 60 boxes containing 600 capsules each (lasting for 100 days in maximum).
   * Surrogate markers/parameters from blood and stool are measured at 0wk and 12wk. Blood samples are collected before the exercise tests. The subjects will bring the samples of their last stool before the exercise tests (at weeks 0 and 12) directly to the exercise physiology laboratory. For blood lactate - in the context of performance diagnostics at weeks 0, 4 and 12 - we collect capillary earlobe blood before, during and until 30 minutes post exercise.
   * Subjects monitor stool appearance via Bristol stool scale/protocol. This is conducted the week before the first exercise test and in the 12th week.
   * Quality of life survey is conducted in the running in period (stress profile)
   * The week before the exercise test it is necessary to adhere to a 4-day diet plan (the last 4 days before the test) and to conduct a 7-day food recording. These sanctions are necessary to match carbohydrate, fat, protein and micronutrient intake and to exclude diet-associated biased lactate kinetics.

   MARKERS/PARAMETERS

   • Performance diagnostics: maximum performance in watt (Pmax), maximum oxygen uptake capacity (VO2max), CO2 exhalation, CO2/O2 ratio, lactate kinetics, maximum lactate, lactate turnpoint 1 (LTP1), lactate turnpoint 2 (LTP2) and anaerobic threshold (ANS), respiratory quotient, EKG for cardiocirculatory innocuousness.
   * Minerals (serum/plasma) and standard blood chemistry: Mg, Ca, Fe, K, Na, Al, Si, P, Cl, ALT, AST, creatinine, ferritin, transferrin, uric acid, vitamin C, free testosterone, SHBG (testosterone transporter), FAI (= free androgen index = Testosterone x 100/SHBG).
   * OS/redox biology (serum/plasma): carbonyl proteins (CP), F2-isoprostanes, total oxidation status (TOS), proteinogenic antioxidant capacity (PAOC), non-proteinogenic antioxidant capacity (NPAOC), DNA strand breaks, glutathione peroxidase 3.
   * Inflammation/immunity (blood/serum/plasma): TNF-alpha, IL-6, IL-8, IL-10, IL-22.
   * Intestinal barrier integrity and endotoxemia: Zonulin (stool), claudin1 and claudin2 (stool), lipopolysaccharides (blood), toll-like receptors (TLR2 and TLR4 from blood), gut profile "basis" (kind and number of colonies, Calprotectin, α1-antitrypsin etc).
   * Body fat determination and distribution via lipometry (non-invasive) at weeks 0 and 14.

   BLOOD SAMPLING

   • Week 0: At rest, after 4wk wash-out and before 1st performance diagnostics
   * Week 12: At rest, after 12wk before 3rd performance diagnostics
   * Capillary blood from earlobe to determine lactate is drawn before, during and after exercise at weeks 0, 4 and 12: at each step of exercise and 3, 6, 9, 12, 15, 20 and 30 min post exercise to evaluated recovery lactate kinetics.

   STOOL SAMPLING
   * Week 0: At rest, after 4 wk wash-out and before 1st performance diagnostics
   * Week 12: At rest, before 3rd performance diagnostics

   PROTOCOLS/QUESTIONNAIRES

   • Stool protocol is conducted the week before 1st and 3rd performance testing

   • Food habits are documented by food recording and the diet plan the last week prior to each exercise test, at weeks 0, 4 and 12
   * Exercise and trainings habits are evaluated by the sport scientist via interview before each performance testing
   * Psycho-social well-being and stress perception are evaluated with the "Quality of Life-BREF" questionnaire (SF36) before the 1st and 3rd performance testing

   PERFORMANCE DIAGNOSTIC (PD) PD is a cycle-steptest-ergometry to performance/watt maximum, lactate maximum and VO2max.. After 3 min rest on the cycle ergometer, subjects start exercise with another 3 min warm up at 60 watt. Then they increase exercise intensity by 15 watt per min (with constant 80 rpm) until exhaustion/VO2max. After reaching exhaustion/VO2max, candidates continue to perform at low intensity (at 30% of Pmax) for further 30 minutes to observe recovery lactate kinetics.

   All tests are supervised by a physician and a sport scientist. Before each test, volunteers are also checked by the physician.

   PD is conducted at:

   • Week 0: 1st performance diagnostics = last selection of candidates (detailed medical check, standard blood chemistry panel)

   • Week 4: 2nd performance diagnostics

   • Week 12: 3rd and last performance diagnostics

   LIPOMETRY
   * Week 0: At rest, after 4wk wash-out and before 1st performance diagnostics
   * Week 12: At rest, after 12wk of supplementation and before 3rd performance diagnostics

   SAMPLE SIZE CALCULATION & RANDOMIZATION Sample size calculation is based on the expectation of an 8% increase in performance capability (in watt) after 4 weeks of treatment with zeolite + dolomite ("PANACEO-SPORT"), compared to placebo (no change). The investigators expect an average Pmax of 345 watt in this trained cohort, a standard deviation of 10%, and chose a power of 80% for this 2-arm design (1:1 distribution of placebo/verum). This calculation revealed a number of 50 subjects. Drawing into account a drop out rate of 10%, we recommend a sample size of 56 subjects, 28 in each group.

   Subjects will be randomized into blocks of 4 (2 verum and 2 placebos in each block) and sequentially numbered (www.randomization.com). To guarantee a balanced distribution in performance capability/VO2max between groups (verum vs. placebo) we will conduct stratification via VO2max rank statistics. The allocation of the capsules/boxes will be conducted after the completed 1st exercise test session. Boxes will be delivered by mail and in 2 tranches (a 7 blocks or 28 subjects), separated by a week. This scheme considers a one week period to check 28 subjects and therefore ensures equal duration of treatment for all candidates.

   STATISTICAL ANALYSES For blood and stool data we will use an univariate, two-factorial analysis of variance (ANOVA). Factors: "treatment" (= placebo vs product) and "time" (= week 0 vs week 12). For lactate and other performance diagnostic parameters we use a three-factorial repeated measures ANOVA with the additional factor "session" (test 1, 2, 3). This statistical test method ensures the consideration of all before-, during- and after- measurements. Further, we will use non-parametric tests, descriptive statistics, and - if indicated - correlation analyses.

ELIGIBILITY:
Inclusion Criteria:

* trained people
* non-smokers
* body fat: 20-30%
* 4wk wash-out 20-50 years old

Exclusion Criteria:

* sedentary people
* smokers
* people not eligible for exercise
* high/low body fat
* people taking supplements
* to young/old people

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of aerobic performance capability between baseline, 4 and 12 weeks | 0, 4, 12 weeks
  Zeolite and Dolomite might influence maximum aerobic performance due to attenuated lactate accumulation in a step test ergometry

SECONDARY OUTCOMES:
Change of lactate concentrations in blood between baseline, 4 and 12 weeks | 0, 4, 12 weeks
  Lactate accumulation and -kinetics is influenced by dietary zeolite and dolomite supplementation

OTHER OUTCOMES:
Change in redox biology between baseline, 4 and 12 weeks | 0, 4, 12 weeks
  Zeolite + dolomite show attenuation of oxidation during and after intense aerobic exercise

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, Prof, Principal Investigator — Green Beat
Locations (1):
- Green Beat, Graz, Austria